CLINICAL TRIAL: NCT04627454
Title: Evaluation the Safety and Effectiveness of Dynamic Cervical Implants (DCI) in Treatment of Single Level Cervical Disc Disease
Brief Title: Dynamic Cervical Implant in Treatment of Cervical Disc Disease
Acronym: DCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fahd Abdel Sabour Ahmed Mohammed, Principal investigator, Resident doctor, neurosurgery department, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DCI in cervical disc disease
Record Dates: First submitted 2020-09-01; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Cervical Disc Disease; Cervical Disc Herniation; Cervical Disc Degeneration
Keywords: Dynamic cervical implant
MeSH Terms: interventions — Diskectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dynamic cervical implant (Experimental): dynamic cervical implant in treatment of cervical disc disease
  Interventions: Procedure: Discectomy and insertion of dynamic cervical implant in cervical disc herniation
- discectomy (Experimental): insertion of dynamic cervical implant post cervical discectomy single level
  Interventions: Procedure: Discectomy and insertion of dynamic cervical implant in cervical disc herniation

INTERVENTIONS:
Procedure: Discectomy and insertion of dynamic cervical implant in cervical disc herniation — The surgical technique included the use of a conventional anterior cervical approach and discectomy and insertion of dynamic cervical implant after discectomy without fixation

SUMMARY:
* Evaluation of outcome of DCI in treatment of cervical disc disease to patients admitted to neurosurgery department, Asyut University Hospitals.
* Give the effective treatment, pain control and can detect the best method could be used.
* Improve the outcome of these patients and decease rate of recurrence and complications.

DETAILED DESCRIPTION:
Anterior cervical decompression and fusion (ACDF) is the traditional method for treating degenerative cervical disc disease, providing satisfactory results in a high proportion of patients. However, stabilization of the treated segment may result in loss of mobility as a functional spinal unit and acceleration of degeneration of the adjacent disc. Re operations may be required to treat complications of fusion, such as recurrent radicular symptoms, non-union, graft collapse, or expulsion. Many previous studies have shown that loss of motion at the fused level is compensated by increased motion at adjacent segments after ACDF, which induces a high rate of degenerative change adjacent to the fused segment. Cervical non-fusion techniques have increasingly been accepted and applied by spine surgeons. As a main component of cervical non-fusion techniques, artificial cervical disc replacement provides good ROM of the cervical spine. Dynamic cervical stabilization with the DCI is a novel treatment approach for cervical disc disease that was initially conceived as a method to combine the potential advantages of fusion and total disc replacement. The first DCI was designed by Matgé in 2002 for treating cervical spondylosis. Paradigm spine introduced the second generation DCIs in 2005. A U-shaped appearance and axial elasticity are two the most significant characteristics. A prospective study by Matgé et al. in 2009 showed that the clinical efficacy was satisfactory after DCI replacement in 102 cases of cervical spondylosis and during a 1-year follow-up; there was neither device migration nor subsidence. The basic concept of the inter-body implant is to maintain a distraction-compression mechanism and so avoid possible collapse of the disc height. This is achieved using the special titanium-alloy DCI, which is bio compatible, available in various sizes, and provided with different foot prints. The U-shaped body provides support and has tooth-like serrations that resist expulsion or retropulsion of the implant when placed into the inter-vertebral space. With the end-plate left intact, osteogenesis and bone fusion are inhibited and no further hetero-topic fusions are supposed to occur. The initial clinical and radio graphic results with the DCI appear promising as an alternative to TDR and ACDF in the treatment of cervical disc disease. It affords maximal neurological improvement, along with maintenance of excellent clinical outcomes. The potential bio-mechanical advantages of DCI include the ability to maintain device-level motion and minimize the development of adjacent-segment disease, while protecting the facet joints from excessive stresses noted with other motion-preserving devices during lateral bending, axial rotation, and extension. The surgical technique included the use of a conventional anterior cervical approach and discectomy. As reported, disc replacement with DCI is a new strategy, in between ACDF & ADR. It is an intermediate solution in the spectrum of management strategies of cervical disc diseases. Immediate dynamic stability with good clinical response and no implant-related morbidity or complications are the main advantages of this implant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with single level cervical disc herniation ( C3 - C7 ).
* Patients with cervical canal stenosis.
* Patients with degenerative disc disease.
* Patient with cervical disc disease not responding to medical treatment.
* Age of the patient: any age.
* Patients fit for surgery.

Exclusion Criteria:

* Patients with multilevel cervical disc herniation.
* Patients with segmental instability.
* Patients with previous cervical spine surgery.
* Patients with cervical kyphosis, active infection or known allergy to titanium.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-11-25 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Change of preoperative neck and radicular pain | Two days post operative
  Pain measurement post op. To evaluate the effectiveness of DCI ( by Oswestry disability index ) that is measured through 10 questions each is. Scored from 0 to 5. A maximum score of 50, then multiply the results by 2 . Scores are stratified into severity: 0-20 minor disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippling bback bain, 81-100 either patients are bed ridden or they are exaggerated their symptoms.
Evaluation the motor power | Three months
  Evaluation patients' motor activity comparing preoperative and postoperative motor power.Assessment of motor function can be graded in patients able to obey commands as follows (right compared to left.

CONTACTS AND LOCATIONS:
Overall Officials: Abdel Hai Moussa Abdel Latif, prof., Study Director — Assiut university hospital, neurosurgery department; Ahmed Elsayed Abo Kresha, prof., Study Director — Assiut university hospital, neurosurgery department; Mohammed Elsayed Mahmoud, Prof., Study Director — Assiut university hospital, neurosurgery department

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/15541695/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/9474724/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/12435970/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/19127159/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/19262984/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/10225797/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/14748566/
- See also: Related Info — https://europepmc.org/article/med/12902946
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/18785525/
- See also: Related Info — https://doi.org/10.3171/foc.2004.17.3.10
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/17355018/
- See also: Related Info — https://thejns.org/downloadpdf/journals/j-neurosurg-spine/22/3/article-p237.pdf
- See also: Related Info — https://www.banglajol.info/index.php/BMRCB/article/download/12884/9251
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/17721713/
- See also: Related Info — https://www.google.com/search?rlz=1C1CHBD_arEG909EG909&sxsrf=ALeKk02OsmpENAj4A5tcvZVyY4KF8Rl3eA:1599003417496&q=18.%09De+Bowes+RM,+Grant+BD,+Bagby+GW,+Butts+MK.+Cervical+vertebral+interbody+fusion+in+the+horse:+a+comparative+study+of+bovine+xenografts+and+allografts+supported+by+stainless+steel+baskets.+Am+J+Vet+Res+1984;+45:+191-9&spell=1&sa=X&ved=2ahUKEwjJ4cb1j8nrAhUO1BoKHbpSBu8QkeECKAB6BAgKECo